CLINICAL TRIAL: NCT04450069
Title: A Phase 1, Open-label, Dose Escalating Study Evaluating the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Clinical Activity of the Combination of CLBR001 and SWI019 in Patients With Relapsed/Refractory B-cell Malignancies
Brief Title: CLBR001 and SWI019 in Patients With Relapsed / Refractory B-cell Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Calibr, a division of Scripps Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CBR-sCAR19-3001
Record Dates: First submitted 2020-06-23; First posted 2020-06-29 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Relapsed/Refractory B-cell Lymphomas; Diffuse Large B Cell Lymphoma (DLBCL); Follicular Lymphoma (FL); Chronic Lymphocytic Leukemia (CLL); Marginal Zone Lymphoma (MZL); Mantle Cell Lymphoma; Small Lymphocytic Lymphoma (SLL); Primary Mediastinal Large B Cell Lymphoma; Transformed Follicular Lymphoma; Waldenstrom Macroglobulinemia; Lymphoplasmacytic Lymphoma; Burkitt Lymphoma
Keywords: CAR-T Cell Therapy; Switchable CAR-T Cell; Autologous Cell Therapy; CD19 Positive Disease; CD19 CAR-T Cell; Blood Cancer; Hematological malignancy; Neoplasms
MeSH Terms: conditions — Lymphoma, B-Cell; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Mantle-Cell; Waldenstrom Macroglobulinemia; Burkitt Lymphoma; Hematologic Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dose Escalation (Experimental): CLBR001 + SWI019 is administered via infusion with ascending dose levels to determine the maximum tolerated dose (MTD) or optimal SWI019 dose (OSD)
  Interventions: Combination Product: CLBR001 and SWI019

INTERVENTIONS:
Combination Product: CLBR001 and SWI019 — Investigational immunotherapy for B cell malignancies

SUMMARY:
CLBR001 + SWI019 is an combination investigational immunotherapy being evaluated as a potential treatment for patients diagnosed with B cell malignancies who are refractory or unresponsive to salvage therapy or who cannot be considered for or have progressed after autologous hematopoietic cell transplantation. This first-in-human study will assess the safety and tolerability of CLBR001 + SWI019 and is designed to determine the maximum tolerated dose (MTD) or optimal SWI019 dose (OSD). Patients will be administered a single infusion of CLBR001 cells followed by cycles of SWI019. The study will also assess the pharmacokinetics and pharmacodynamics of CLBR001 + SWI019.

DETAILED DESCRIPTION:
CLBR001 + SWI019 is a two-component therapy comprising an autologous chimeric antigen receptor T (CAR-T) cell product (CLBR001, the switchable CAR-T cell (sCAR-T)) and an anti-CD19 (cluster of differentiation antigen 19) antibody (SWI019, the switch, a biologic). In combination, SWI019 acts as an adapter molecule that controls the activity of the CLBR001 CAR-T cell product.

ELIGIBILITY:
Inclusion Criteria:

* Patients with relapsed / refractory previously treated B cell malignancies (according to the World Health Organization classification; 2017)
* Patients must have received adequate prior therapy including at least two lines of prior therapies including anthracycline or bendamustine-containing chemotherapy, anti-CD20 (cluster of differentiation antigen 20) therapies and/or Brutton's tyrosine kinase (BTK) inhibitors
* Patients treated with prior CD19 targeted molecules (e.g., Blincyto) must have confirmed CD19+ disease
* Patients must be ineligible for allogeneic stem cell transplant (SCT)
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0 or 1
* Estimated life expectancy of ≥ 12 weeks from the first day of SWI019 dose administered
* Willing to undergo pre- and post-treatment core needle biopsy
* Adequate hematological, renal, pulmonary, cardiac, and liver function
* Resolved adverse events of any prior therapy to either baseline or CTCAE Grade ≤1
* Women of childbearing potential, a negative pregnancy test and must agree to practice effective birth control
* Men sexually active with female partners of child bearing potential must agree to practice effective contraception
* Willing and able to comply with scheduled visits, treatment plan, laboratory tests and other procedures

Exclusion Criteria:

* Patients diagnosed with certain disease histologies including pediatric lymphomas/leukemias, monoclonal gammopathy of undetermined significance (MGUS), T-cell histiocyte large B cell lymphoma
* Pregnant or lactating women
* Active bacterial, viral, and fungal infections
* History of allogeneic stem cell transplantation
* Treatment with any prior lentiviral or retroviral based CAR-T
* Patients receiving live (attenuated) vaccines within 4 weeks of screening visit or need for live vaccine on study
* Patients with known active central nervous system (CNS) disease. Patients with prior CNS disease that has been effectively treated may be eligible
* History of Class III or IV New York Heart Association (NYHA) heart failure, myocardial infarction, unstable angina or other significant cardiac disease within 6 months of screening
* Involvement of cardiac tissue by lymphoma
* Uncontrolled autoimmune hemolytic anemia or idiopathic thrombocytopenic purpura (ITP)
* HIV-1 and HIV-2 antibody positive patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2020-08-14 (Actual); Primary Completion 2024-05-06 (Actual); Study Completion 2024-05-06 (Actual)

PRIMARY OUTCOMES:
Frequency, relatedness, severity and duration of treatment emergent and treatment related adverse events | 35 days
  To determine the frequency, relatedness, severity and duration of treatment emergent and treatment related adverse events
Number of first cycle dose limiting toxicities (DLT) as assessed by Common Terminology Criteria for Adverse Events (CTCAE) | up to 1 year
  Based on the number of first cycle dose limiting toxicities (DLT) as assessed by CTCAE to determine maximum tolerated dose (MTD)

SECONDARY OUTCOMES:
Maximum drug concentration (Cmax) of SWI019 | up to Day 35
  To determine the maximum concentration of SWI019 in a patient's peripheral blood
Area under the curve (AUC) of SWI019 | up to Day 35
  To quantify the cumulative amount of SWI019 in a patient's peripheral blood over time
Time to reach Cmax (Tmax) of SWI019 | up to Day 35
  To identify the time point when the concentration of SWI019 reaches maximum in a patient's peripheral blood
Clearance (CL) of SWI019 | up to Day 35
  To determine the clearance factor of SWI019 in a patient's peripheral blood
Apparent elimination half-life (t1/2) of SWI019 | up to Day 35
  To identify the time point when the concentration of SWI019 reaches half of maximum in a patient's peripheral blood
Quantification of CLBR001 cells in peripheral blood | up to 1 year
  To quantify CLBR001 in a patient's peripheral blood at different time points
Phenotype of CLBR001 in peripheral blood and/or tumor/bone marrow biopsies | up to 1 year
  To evaluate the phenotype of CLBR001 in a patient's peripheral blood at different time points by flow cytometry
Immunogenic response to CLBR001 | up to 1 year
  To evaluate the anti-drug antibodies in response to CLBR001 administration in a patient's peripheral blood
Immunogenic response to SWI019 | up to 1 year
  To evaluate the anti-drug antibodies in response to SWI019 administration in a patient's peripheral blood
Serum cytokine concentrations | up to 1 year
  To measure the cytokine levels (e.g. TNFa, IL-6, IL-1, IL-2, etc.) in a patient's peripheral blood at different time points
Overall (best) objective response by the Response Evaluation Criteria in Lymphoma (RECIL) and Lugano criteria | up to 1 year
  To determine the overall (best) objective anti-cancer response by RECIL and Lugano criteria
Duration of response (DOR) | up to 1 year
  To evaluate the duration of anti-cancer response after CLBR001 and SWI019 administration
Progression free survival (PFS) | up to 1 year
  To evaluate the duration of patient's progression-free survival
Overall survival (OS) | up to 1 year
  To evaluate the overall duration of patient's survival

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - City of Hope National Medical Center, Duarte, California
  - University of California at San Diego, San Diego, California
  - University of Chicago, Chicago, Illinois
  - Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota
  - Weill Cornell Medical College - New York Presbyterian Hospital, New York, New York
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - Sarah Cannon Research Institute - Tennessee Oncology, Nashville, Tennessee
  - Sarah Cannon Research Institute - Texas Transplant Institute, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rodgers DT, Mazagova M, Hampton EN, Cao Y, Ramadoss NS, Hardy IR, Schulman A, Du J, Wang F, Singer O, Ma J, Nunez V, Shen J, Woods AK, Wright TM, Schultz PG, Kim CH, Young TS. Switch-mediated activation and retargeting of CAR-T cells for B-cell malignancies. Proc Natl Acad Sci U S A. 2016 Jan 26;113(4):E459-68. doi: 10.1073/pnas.1524155113. Epub 2016 Jan 12. PMID 26759369
- [Background] Viaud S, Ma JSY, Hardy IR, Hampton EN, Benish B, Sherwood L, Nunez V, Ackerman CJ, Khialeeva E, Weglarz M, Lee SC, Woods AK, Young TS. Switchable control over in vivo CAR T expansion, B cell depletion, and induction of memory. Proc Natl Acad Sci U S A. 2018 Nov 13;115(46):E10898-E10906. doi: 10.1073/pnas.1810060115. Epub 2018 Oct 29. PMID 30373813
- [Derived] Ernst M, Oeser A, Besiroglu B, Caro-Valenzuela J, Abd El Aziz M, Monsef I, Borchmann P, Estcourt LJ, Skoetz N, Goldkuhle M. Chimeric antigen receptor (CAR) T-cell therapy for people with relapsed or refractory diffuse large B-cell lymphoma. Cochrane Database Syst Rev. 2021 Sep 13;9(9):CD013365. doi: 10.1002/14651858.CD013365.pub2. PMID 34515338